CLINICAL TRIAL: NCT05180279
Title: The Impact of Circadian Misalignment on Colonic Barrier Homeostasis in Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ali Keshavarzian, Principal Investigator, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19051402; R01DK124280 (NIH)
Record Dates: First submitted 2021-12-14; First posted 2022-01-06 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis
Keywords: Circadian Rhythms
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: 40 human subjects will be recruited into this proposed study: 20 Healthy Controls and 20 UC subjects with left sided inactive disease. Patients will be matched with Health Controls. Patients will have two study visits: the first is the initial in-clinic screening and the second is the 7-day sleep lab intervention. There will be no follow-up after the lab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Lab (Experimental)
  Interventions: Behavioral: 7-day sleep lab

INTERVENTIONS:
Behavioral: 7-day sleep lab — Patients will stay in 7-day sleep lab where light exposure, diet, and activity will be closely monitored. They will have two unprepped flexible sigmoidoscopies with rectal biopsy collection and stool collection. Cycles will be shifted by 12h once on Day 3 of sleep lab and be discharged after an 8 hour sleep session on Day 7.

SUMMARY:
The purpose of this study is to investigate if circadian malalignment (unusual sleeping patterns), such as night shifts (sleeping during the day and being awake during the night time), worsens the inflammation of the gut. We hope to look at patients with Ulcerative Colitis and Healthy Controls.

ELIGIBILITY:
Inclusion Criteria:

UC patients:

* M/F, 18-50 y/o
* Inactive Disease (Mayo Score ≤ 2)
* Stable medications with no disease flares for the > 3 months
* Left-sided UC (Montreal E1 or E2)
* Normal psychological evaluation and negative drug screen (See Below)

Healthy Controls:

* M/F, 18-50 y/o, age ± 3y sex, race, and BMI match with UC subject
* No clinical evidence of any medical illness
* Normal psychological evaluation and negative drug screen (See Below)

Exclusion Criteria:

UC patients:

* Patients with other forms of colitis such as Crohn's disease (CD) or indeterminate colitis
* Patient with active UC (Mayo > 2)
* Pancolonic UC (colitis past the splenic flexure, Montreal E3))
* Use of biologic or immunomodulatory medications (i.e. Infliximab, Adalimumab, azathioprine, Vedolizumab, methotrexate, etc.)
* Gastrointestinal surgery
* Other GI diseases or systemic diseases (cardiac, renal failure, cirrhosis)
* Shift work in the last 6 months
* Antibiotic use within last 12 weeks
* Patients who have used anti-diarrheal agents such as Lomotil or Imodium within 3 days of the study
* Prednisone use the last 30 days
* Significant Depression (score ≥ 14 BDI)
* Significant Anxiety (score ≥ 40 STAI)
* Use of probiotic supplement in last 4 weeks except yogurt.
* Intentional change in diet.
* Chronic use of NSAIDS. A washout period of 3 weeks is needed before the subject could be enrolled into the study. Low dose aspirin is allowed.
* Chronic Alcohol use. A washout period of 3 weeks is needed before the subject could be enrolled into the study.
* Have children under 6 months

Healthy Controls:

* History of drug abuse, gastrointestinal (GI) surgery, GI diseases, or systemic diseases such as renal (creatinine>1.2 mg/dl), liver, cardiac, or diabetes (Hgb-A1c>8%)
* Antibiotic use within last 12 weeks
* Shift work in the last 6 months
* Use of probiotic supplement except yogurt in last 4 weeks.
* Atypical American diet with daily fiber ≥ 16 grams or daily saturated fat ≤ 11 grams by Food Frequency Questionnaire
* Chronic use of NSAIDS. A washout period of 3 weeks is needed before the subject could be enrolled into the study.
* Chronic Alcohol use. A washout period of 3 weeks is needed before the subject could be enrolled into the study.
* Significant Depression (score ≥ 14 BDI)
* Significant Anxiety (score ≥ 40 STAI)
* Regular use of medications that affect intestinal permeability, intestinal motility and/or endogenous melatonin including metoclopramide, NSAIDs, antibiotics, beta blocker, psychotropic medication, hypnotics and exogenous melatonin products during 4 weeks prior to the study
* People who crossed more than 2 time zones in the previous month
* Inability to sign an informed consent form.
* Have children under 6 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Control: 7-day sleep lab: Healthy Control participants (no ulcerative Colitis) will stay in 7-day sleep lab where light exposure, diet, and activity will be closely monitored. Participants at baseline will not have a misaligned circadian rhythm. They will have two unprepped flexible sigmoidoscopies with rectal biopsy collection and stool collection at baseline and after misalignment. Cycles will be shifted by 12h once on Day 3 of sleep lab and be discharged after an 8-hour sleep session on Day 7.
- Ulcerative Colitis: 7-day sleep lab: Participants with ulcerative colitis will stay in 7-day sleep lab where light exposure, diet, and activity will be closely monitored. Participants at baseline will not have a misaligned circadian rhythm. They will have two unprepped flexible sigmoidoscopies with rectal biopsy collection and stool collection at baseline and after misalignment. Cycles will be shifted by 12h once on Day 3 of sleep lab and be discharged after an 8-hour sleep session on Day 7
Period: Overall Study
Arm/Group | Healthy Control | Ulcerative Colitis
Started | 9 | 10
Completed | 7 | 10
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Control: 7-day sleep lab: Healthy Control participants (no ulcerative colitis) will stay in 7-day sleep lab where light exposure, diet, and activity will be closely monitored. Participants at baseline will not have a misaligned circadian rhythm. They will have two unprepped flexible sigmoidoscopies with rectal biopsy collection and stool collection at baseline and after misalignment. Cycles will be shifted by 12h once on Day 3 of sleep lab and be discharged after an 8 hour sleep session on Day 7.
- Ulcerative Colitis: 7-day sleep lab: Participants with ulcerative colitis will stay in 7-day sleep lab where light exposure, diet, and activity will be closely monitored. Participants at baseline will not have a misaligned circadian rhythm. They will have two unprepped flexible sigmoidoscopies with rectal biopsy collection and stool collection at baseline and after misalignment. Cycles will be shifted by 12h once on Day 3 of sleep lab and be discharged after an 8 hour sleep session on Day 7.
- Total: Total of all reporting groups
Arm/Group | Healthy Control | Ulcerative Colitis | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 10 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 32 [21 to 54] | 23.5 [18 to 35] | 24 [18 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 3 | 6 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2 | 4 | 6
  African American | 3 | 0 | 3
  Hispanic or Latino | 2 | 4 | 6
  African | 0 | 1 | 1
  Asian | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Dim Light Melatonin Onset (DLMO) From Baseline (Aligned) to Circadian Misalignment Misalignment
Description: Amount of time between dim light melatonin onset (DLMO) to sleep onset. The hours reported for this outcome measure equates the time of the day the participant fell asleep
Time Frame: Blood is drawn every hour over 8 hours to measure plasma melatonin in dim light < 5 lux in Aligned Circadian Rhythms, and blood is drawn every hour for 12 hours under dim light in Misaligned Circadian rhythms.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Healthy Control: 7-day sleep lab: Healthy control participants (no ulcerative colitis) will stay in 7-day sleep lab where light exposure, diet, and activity will be closely monitored. Participants at baseline will not have a misaligned circadian rhythm. They will have two unprepped flexible sigmoidoscopies with rectal biopsy collection and stool collection. Cycles will be shifted by 12 hours once on Day 3 of sleep lab and be discharged after an 8-hour sleep session on Day 7.
- Ulcerative Colitis: 7-day sleep lab: Participants with ulcerative colitis will stay in 7-day sleep lab where light exposure, diet, and activity will be closely monitored. Participants at baseline will not a have a misaligned circadian rhythm. They will have two unprepped flexible sigmoidoscopies with rectal biopsy collection and stool collection. Cycles will be shifted by 12h once on Day 3 of sleep lab and be discharged after an 8 hour sleep session on Day 7
Arm/Group | Healthy Control | Ulcerative Colitis
Number analyzed (Participants) | 7 | 10
hours
  Baseline Aligned Circadian Rhythm | 20.72 (0.52) | 20.45 (1.08)
  Misaligned Circadian Rhythm | 23.05 (0.48) | 22.65 (1.88)

2. Primary Outcome: Change in Intestinal Permeability From Baseline (Aligned Circadian Rhythms) to Circadian Misalignment
Description: Intestinal permeability is assessed through spectrophotometric measurements of sucralose, sucrose, maltose and lactulose concentrations in urine following ingestion of a sugar cocktail.
Time Frame: 24 hour urine collection beginning at baseline and 24 hour urine collection at circadian misalignment, an average of 3 days from baseline to circadian misalignment
Measure: Mean (Standard Deviation); unit: % excretion of oral dose 12-24 hr urinar
Groups:
- Healthy Control: 7-day sleep lab: Healthy Control participants will stay in 7-day sleep lab where light exposure, diet, and activity will be closely monitored. Participants at baseline will not have a misaligned circadian rhythm. They will have two unprepped flexible sigmoidoscopies with rectal biopsy collection and stool collection at baseline and after misalignment. Cycles will be shifted by 12h once on Day 3 of sleep lab and be discharged after an 8 hour sleep session on Day 7.
- Ulcerative Colitis: 7-day sleep lab: Patients will stay in 7-day sleep lab where light exposure, diet, and activity will be closely monitored. Participants at baseline will not have a misaligned circadian rhythm. They will have two unprepped flexible sigmoidoscopies with rectal biopsy collection and stool collection. Cycles will be shifted by 12h once on Day 3 of sleep lab and be discharged after an 8 hour sleep session on Day 7
Arm/Group | Healthy Control | Ulcerative Colitis
Number analyzed (Participants) | 7 | 10
% excretion of oral dose 12-24 hr urinar
  Baseline Aligned Circadian Rhythm | 0.053 (0.040) | 0.141 (0.065)
  Misaligned Circadian Rhythm | 0.088 (0.053) | 0.184 (0.111)

3. Secondary Outcome: Change in 24 Hour Urinary Melatonin Concentrations From Baseline (Aligned Circadian Rhythms) to Circadian Misalignment
Description: Spectrophotometry
Time Frame: 24 hour urine collection at baseline and 24 hour urine collection at circadian misalignment circadian
Reporting Status: Not Posted

4. Secondary Outcome: Change in Mayo Score From Baseline (Aligned Circadian Rhythms) to Circadian Misalignment
Description: Within the endoscopic component of the Mayo Score, a score of 0 is given for normal mucosa or inactive UC, while a score of 1 is given for mild disease with evidence of mild friability, reduced vascular pattern, and mucosal erythema.
Time Frame: 30 minute flexible sigmoidoscopy at Baseline and 30 minute flexible sigmoidoscopy at Circadian Misalignment
Reporting Status: Not Posted

5. Secondary Outcome: Change in Stool Calprotectin From Baseline (Aligned Circadian Rhythms) to Circadian Misalignment
Description: Calprotectin is a sensitive marker for inflammation in the gastrointestinal tract. Measured through enzyme linked immunosorbent assay for calprotectin in stool extract.
Time Frame: 10 minute stool collection conducted at baseline circadian rhythm and at circadian misalignment.
Reporting Status: Not Posted

6. Secondary Outcome: Change in Concentration of Serum Cytokine Markers of Inflammation From Baseline (Aligned Circadian Rhythms) to Circadian Misalignment
Description: Enzyme linked immunosorbent assay
Time Frame: Blood is drawn every two hours over a 24 hour period at baseline (12 draws), and blood is drawn every two hours over a 24 hour period at circadian misalignment
Reporting Status: Not Posted

7. Secondary Outcome: Changes in Clock Gene Expression in Peripheral Blood Mononuclear Cells From Baseline (Aligned Circadian Rhythms) to Circadian Misalignment
Description: RNA Sequencing
Time Frame: as for outcome 6
Reporting Status: Not Posted

8. Secondary Outcome: Changes in Gene Expression of Colonic Tissue Biopsies From Baseline (Aligned Circadian Rhythms) to Circadian Misalignment
Description: Tissue biopsies collected during flexible sigmoidoscopy conducted at Baseline Circadian Rhythm and at Circadian Misalignment. Assessed through histology and RNA Sequencing
Time Frame: 30 minute flexible sigmoidoscopy at Baseline and 30 minute flexible sigmoidoscopy at Circadian Misalignment
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Diet
Description: Vioscreen Food Frequency Questionnaire (FFQ). Total of 19 measured food components. Vioscreen captures comprehensive dietary behaviors in just 30 minutes. It is a unique dietary questionnaire, management and analysis system that efficiently gathers and manages data that immediately identifies dietary "habits" and counsel for lifestyle changes.
Time Frame: Once before sleep lab
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Single Day Food Recall
Description: Automated Self-Administered 24-Hour Recall (ASA24) Dietary Assessment. Total nutrients from all supplements reported in a given day.
Time Frame: Once before sleep lab
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Chronotype
Description: The Munich ChronoType Questionnaire (MCTQ) uses a self-rated scale to assess individual phase of entrainment on work and work-free days; it is a tool to collect primary sleep times, such as bed- and rise-times, plus the clock time of becoming fully awake as well as sleep latency and inertia, in addition to other time points.
Time Frame: Screening
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Beck Depression Inventory
Description: The Beck Depression Inventory (BDI, BDI-II), created by Dr. Aaron T. Beck, is a 21-question multiple-choice self-report inventory, one of the most widely used instruments for measuring the severity of depression.
Time Frame: 3 Weeks prior to circadian lab assessments
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Pittsburgh Sleep Quality Index
Description: The following questions relate to your usual sleep habits during the past month only.
Time Frame: 3 Weeks prior to circadian lab assessments
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 days
Groups:
- Healthy Controls; Ulcerative Colitis: 7-day sleep lab: Patients will stay in 7-day sleep lab where light exposure, diet, and activity will be closely monitored. They will have two unprepped flexible sigmoidoscopies with rectal biopsy collection and stool collection. Cycles will be shifted by 12h once on Day 3 of sleep lab and be discharged after an 8 hour sleep session on Day 7.
Arm/Group | Healthy Controls | Ulcerative Colitis
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 0/7 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT05180279/Prot_SAP_003.pdf
  • Informed Consent Form (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT05180279/ICF_002.pdf